CLINICAL TRIAL: NCT07156149
Title: Fabhalta Capsules Specified Drug-use Survey(C3 Glomerulopathy, CLNP023B11401)
Brief Title: Fabhalta Capsules Specified Drug-use Survey
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLNP023B11401
Record Dates: First submitted 2025-09-03; First posted 2025-09-05 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: C3 Glomerulopathy
Keywords: C3 glomerulopathy; C3G; Fabhalta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (1):
- iptacopan: patients administered iptacopan in clinical practice

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of Fabhalta in patients with C3 glomerulopathy in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have used Fabhalta for C3 glomerulopathy (including patients with recurrent C3 glomerulopathy post renal transplant).

Exclusion Criteria:

* Use of iptacopan for an indication not yet approved under the Clinical Trials Act or GCP (e.g., patient-requested medical treatment, investigator-initiated clinical trial)

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who received Fabhalta.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with infections | 360 Days
  Number of patients with infections and type of infections (meningococcal infection, pneumococcal infection, Haemophilus influenzae infection, and other infections based on the causative bacteria) as adverse events/adverse reactions during the treatment period

SECONDARY OUTCOMES:
Incidence of adverse events and adverse reactions | 360 Days
  Incidence of adverse events and adverse reactions that occurred during the treatment period
Changes in UPCR | Baseline, 360 Days
  Changes in UPCR from baseline to Day 360 and from baseline to 360 days
Changes in eGFR | Baseline, 360 Days
  Changes in eGFR from baseline to Day 360 and from baseline to 360 days
Proportion of patients achieving the composite renal endpoint at the final assessment. | 360 Days
  The composite renal endpoint requirement will be met if the following criteria are met: (1) stable or improved eGFR relative to start of treatment (≤ 15% reduction in eGFR) and (2) decrease in UPCR by ≥ 50% relative to start of treatment. Initiation of a complement pathway modulator, initiation/intensification of corticosteroids or immunosuppressants (e.g., MMF) for C3 glomerulopathy, or renal replacement therapy will be determined as failure of the endpoint.
Changes in blood urea nitrogen (BUN) | 360 Days
  Changes in blood urea nitrogen over the course of treatment
Changes in serum albumin | 360 Days
  Changes in serum albumin over the course of treatment
Changes in serum creatinine | 360 Days
  Changes in serum creatinine over the course of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- Japan (10):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Komatsu, Ishikawa-ken
  - Novartis Investigative Site, Tsu, Mie-ken
  - Novartis Investigative Site, Takatsuki, Osaka
  - Novartis Investigative Site, Kusatsu, Shiga
  - Novartis Investigative Site, Ohtsu, Shiga
  - Novartis Investigative Site, Fuchū, Tokyo
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Wakayama

IPD SHARING:
Plan to Share IPD: No